CLINICAL TRIAL: NCT02658708
Title: Bright Light on Fatigue in Women Being Treated for Breast Cancer: A Pilot Study
Brief Title: Bright Light on Fatigue in Women Being Treated for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201503075
Record Dates: First submitted 2016-01-06; First posted 2016-01-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Breast Neoplasms; Breast Cancer; Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Bright blue-green light (Experimental): Complete the MEQ at screening, the day before 2nd cycle of chemo, and on the day of 3rd cycle of chemo, -21 day light intervention at home for 30 min once a day during 2nd cycle of chemo, Scores of ≤41 (evening types) on MEQ will have light delivered within 30 minutes of waking for 21 consecutive mornings. Score of ≥59 (morning types) on MEQ will have light delivered between 1900-2000 hours for 21 consecutive evenings. Light therapy will be self-administered using a light visor cap. On 2 randomly selected days ambient light will be recorded continuously during waking hours using a digital foot candle datalogging light meter, Continuous ambulatory PSG for 24 hours at the participant's home before and after the light intervention, Complete the fatigue and sleep log on a daily basis and two visual analog scales (VAS) (diurnal fatigue and daytime sleepiness) within half an hour upon awakening, at 1200 hours, 1600 hours, 2000 hours, and within half an hour before going to bed
  Interventions: Other: Bright blue-green light using light visor cap; Other: European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire; Other: Epworth Sleepiness Scale; Other: Pittsburgh Sleep Quality Index; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue; Diagnostic Test: Digital foot candle datalogging light meter (Extech Instrument, Model SDL400); Diagnostic Test: Polysomnography (Easy Ambulatory 2 Cadwell, Kennewick, WA); Other: Horne-Ostberg Morningness-Eveningness Questionnaire; Other: Daily Fatigue and Sleep Log
- Arm 2: Dim red light (Active Comparator): Complete the MEQ at screening, the day before 2nd cycle of chemo, and on the day of 3rd cycle of chemo, 21 day light intervention at home for 30 min once a day during 2nd cycle of chemo, Scores of ≤41 (evening types) on MEQ will have light delivered within 30 minutes of waking for 21 consecutive mornings. Score of ≥59 (morning types) on MEQ will have light delivered between 1900-2000 hours for 21 consecutive evenings. Light therapy will be self-administered using a light visor cap. On 2 days randomly selected days ambient light will be recorded continuously during waking hours using a digital foot candle datalogging light meter, Continuous ambulatory PSG for 24 hours at the participant's home before and after the light intervention, Complete the fatigue and sleep log on a daily basis and two visual analog scales (VAS) (diurnal fatigue and daytime sleepiness) within half an hour upon awakening, at 1200 hours, 1600 hours, 2000 hours, and within half an hour before going to bed
  Interventions: Other: Dim red light using light visor cap; Other: European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire; Other: Epworth Sleepiness Scale; Other: Pittsburgh Sleep Quality Index; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue; Diagnostic Test: Digital foot candle datalogging light meter (Extech Instrument, Model SDL400); Diagnostic Test: Polysomnography (Easy Ambulatory 2 Cadwell, Kennewick, WA); Other: Horne-Ostberg Morningness-Eveningness Questionnaire; Other: Daily Fatigue and Sleep Log

INTERVENTIONS:
Other: Bright blue-green light using light visor cap
  Arms: Arm 1: Bright blue-green light
Other: Dim red light using light visor cap
  Arms: Arm 2: Dim red light
Other: European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire — -Consists of 30 items with a 4-point rating scale (1=not at all to 4=very much) measuring functioning, symptom intensity, and global health status/quality of life
  Other Names: EORCT QLQ C-30
Other: Epworth Sleepiness Scale — -Consists of 8 common daily activities with a 4-point rating scale (0=would never doze to 3=a high chance of dozing) measuring usual daytime sleepiness over a recent time period
  Other Names: ESS
Other: Pittsburgh Sleep Quality Index — -Contains 19 self-report items measuring sleep quality, latency, duration, efficiency, disturbance, medication use, and daytime dysfunction. Each item is rated on a 0-3 rating scale. The global PSQI score ranges 0-21, with higher scores indicating more severe sleep disturbance
  Other Names: PSQI
Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance — -Consists of 8 items with 5-point rating scales measuring overall sleep and sleep-related impairments. Higher scores indicate worse sleep disturbances
Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue — -Consists of 8 items with a 5-point rating scale (1=not at all to 5 =very much) measuring fatigue experience and fatigue impact. Higher scores indicate worse fatigue.
Diagnostic Test: Digital foot candle datalogging light meter (Extech Instrument, Model SDL400) — -The light-weight light sensor is approximately 2 inches in diameter and comes with a clip and strap that makes it comfortable to wear just below the neck.
Diagnostic Test: Polysomnography (Easy Ambulatory 2 Cadwell, Kennewick, WA) — -A standard sleep montage of electroencephalography following the 10/20 procedure for electrode placement, left and right electrooculography referenced to the opposite mastoid and mentalis electromyography will be followed
  Other Names: PSG
Other: Horne-Ostberg Morningness-Eveningness Questionnaire
  Other Names: MEQ
Other: Daily Fatigue and Sleep Log — * Two visual analog scales (VAS) for diurnal fatigue and daytime sleepiness
  * Two 0-10 point rating scales (average and worst fatigue levels in 24 hours)

SUMMARY:
This proposed study will examine feasibility and implement therapeutic bright light that is tailored to the individual's circadian typology to estimate its therapeutic effects on sleep/wake patterns and fatigue in breast cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Newly diagnosed with stage I-III breast cancer
* Scheduled to receive 21-day cycles of intravenous chemotherapy
* Experiencing disrupted sleep (determined by Pittsburgh Sleep Quality Index)
* Morning or evening types (determined by Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ)
* Sighted
* Mentally competent to consent
* Able to under English

Exclusion Criteria:

* Concurrent malignancy
* Undergoing other cancer treatments
* Engage in shift work or travel across more than 3 time zones within 2 weeks prior to study
* Known history of seasonal affective disorder or substance abuse
* Current diagnosis of major Axis I psychiatric disorders, neurological impairments, or muscular dystrophies
* Regularly use steroid or other immunosuppressive medications
* Take prescribed sedative hypnotics or sleep medications because these conditions may affect fatigue and/or sleep/wake patterns.
* Have eye conditions (glaucoma or retinal disease), problems triggered by bright light (e.g. migraine), or take photosensitizing medications (e.g. some porphyrin drugs, antipsychotics, antiarrhythmic agents)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing a bright light intervention as measured by estimating completion of scheduled PSG recording | Through completion of study (approximately 50 days)
  -Feasibility of the procedures will be assessed by descriptive analysis
Effect of bright light on fatigue as measured by PROMIS-Cancer Fatigue | Through completion of study (approximately 50 days)
Effect of bright light on fatigue as measured by VAS (diurnal fatigue) in Daily Fatigue and Sleep Log | Through of completion of study (approximately 43 days)
Effect of bright light on sleep patterns as measured by PSG | Through completion of study (approximately 50 days)
Effect of bright light on sleep patterns as measured by PROMIS-Sleep Disturbance | Through of completion of study (approximately 43 days)
Effect of bight light on sleep patterns as measured by PSQI | Through completion of study (approximately 50 days)
Effect of bright light on wake patterns as measured by PSG | Through completion of study (approximately 50 days)
Effect of bright light on wake patterns as measured by ESS | Through completion of study (approximately 50 days)
Effect of bright light on wake patterns as measured by VAS (daytime sleepiness) in Daily Fatigue and Sleep Log | Through completion of study (approximately 50 days)
Effect of bright light on quality of life as measured by EORCT QLQ C-30 | Through completion of study (approximately 50 days)
Feasibility of implementing a bright light intervention as measured by completion rates of self-report forms | Through completion of study (approximately 50 days)
  -Feasibility of the procedures will be assessed by descriptive analysis

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Shiuann Wu, Ph.D., R.N., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu HS, Davis JE, Chen L. Bright light shows promise in improving sleep, depression, and quality of life in women with breast cancer during chemotherapy: findings of a pilot study. Chronobiol Int. 2021 May;38(5):694-704. doi: 10.1080/07420528.2021.1871914. Epub 2021 Jan 21. PMID 33478260
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu